CLINICAL TRIAL: NCT00632970
Title: A Multi-Center Comparison of Raltegravir to Lopinavir/Ritonavir, Both in Combination With Truvada, in HIV-Infected Individuals Naive to Antiretroviral Therapy
Brief Title: Raltegravir vs. Lopinavir/Ritonavir, Both in Combination With Truvada, in HIV+ Treatment Naive Individuals
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no patients completed
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Gary Simon, Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS001
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
Keywords: Raltegravir; Lopinavir
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Lopinavir; lopinavir-ritonavir drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir plus Truvada (Experimental): Raltegravir (400mg), 1 tablet, administered twice daily (BID) and Truvada (Emtricitabine/Tenofovir disoproxil fumarate) (200mg/300mg), 1 tablet administered once daily (QD)
  Interventions: Drug: Raltegravir; Drug: Truvada
- Lopinavir/Ritonavir plus Truvada (Active Comparator): Lopinavir/Ritonavir (400mg/100mg) (Kaletra), 2 tablets administered twice daily (BID) and Truvada (Emtricitabine/Tenofovir disoproxil fumarate) (200mg/300mg), 1 tablet administered once daily (QD)
  Interventions: Drug: Lopinavir/Ritonavir; Drug: Truvada

INTERVENTIONS:
Drug: Raltegravir — 1, 400mg tablet twice a day, with Truvada 1 tablet once a day
  Other Names: Isentress
  Arms: Raltegravir plus Truvada
Drug: Lopinavir/Ritonavir — 2 tablets twice a day, with Truvada 1 tablet once a day
  Other Names: Kaletra
  Arms: Lopinavir/Ritonavir plus Truvada
Drug: Truvada — 1 tablet, once a day, with either Raltegravir (Isentress) or Lopinavir/Ritonavir(Kaletra)
  Other Names: Emtricitabine/Tenofovir disoproxil fumarate

SUMMARY:
This program is designed to study the efficacy, safety, lipid effects and tolerability of raltegravir compared to lopinavir/ritonavir, in patients with HIV-I infection who have not received prior antiretroviral therapy. All patients will receive concomitant therapy with Truvada.

DETAILED DESCRIPTION:
It is hypothesized that (1) the raltegravir regimen will have similar efficacy in terms of both viral suppression as well as increases in CD4 cell counts and (2) raltegravir will have significantly less impact on plasma lipids, lipoproteins and lipoproteins subtypes, compared with lopinavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV infection confirmed by western blot or HIV RNA.
2. At least 18 years of age.
3. Less than 1 week of prior antiretroviral therapy.
4. In the opinion of the investigator, patients should be clinically stable. Patients may be on chronic suppressive therapy for opportunistic infections such as MAC or CMV.
5. Patients who are of reproductive potential agree to use an acceptable method of birth control throughout the study. Acceptable methods include an intrauterine device (IUD), diaphragm with spermicide, condoms, or abstinence.
6. HIV RNA > 5000 copies/ml. No restriction on CD4 cell count.
7. A negative urine pregnancy test on the day of initiation of therapy.

Exclusion Criteria:

1. Prior treatment with >1week of antiretroviral therapy.
2. Patient requires or is anticipated to require any of the prohibited medications noted in the protocol.
3. HIV RNA < 5000 prior to receiving therapy.
4. Baseline resistance to any of the study regimen drugs on genotype testing.
5. Patients with acute hepatitis due to any cause or clinically significant chronic liver disease.
6. Patient with severe renal insufficiency defined as a calculated creatinine clearance at time of screening <30mL/min, based on the Cockcroft-Gault equation which is as follows (and 0.85X this value for females): Clcr(mL/min) = (l40-age) x weight (in kg)72 x serum creatinine (mg/dL).
7. Patient has a condition (including but not limited to alcohol or other substance abuse) which in the opinion of the investigator would interfere with patient compliance or safety.
8. A female patient who is pregnant, breast-feeding, or expecting to conceive or donate eggs during the study; or a male patient who is planning to impregnate or provide sperm donation during the study is excluded.
9. Inability to obtain signed informed consent from a patient age 18 or older.
10. Patient has significant hypersensitivity or other contraindication to any of the components of the study drug.
11. Patients who should be treated for hyperlipidemia as per NCEPIII guidelines and patients who are currently receiving lipid-lowering therapy are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Simon, MD, PhD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Findings not relevant

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: Patients with HIV infection randomized to receive raltegravir with truvada
- Lopinavir/Ritonavir: Patients with HIV infection randomized to receive lopinavir/ritonavir with truvada
Period: Overall Study
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Raltegravir: Raltegravir: 1 400mg tablet twice a day
- Lopinavir/Ritonavir: Lopinavir/Ritonavir: 2 tablets twice a day
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Lopinavir/Ritonavir | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
HIV seropositive with viral load < 10,000 [Number; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in CD4 Cell Counts
Time Frame: 24 and 48 weeks
Measure: Mean (Full Range); unit: cells/mm^3
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Number analyzed (Participants) | 3 | 3
cells/mm^3 | 50 [10 to 150] | 50 [20 to 120]

2. Secondary Outcome: Change is Plasma Lipids, Lipoproteins and Lipoprotein Subtypes.
Time Frame: 24 weeks
Population: Data can not be reported because the samples were never analyzed and therefore no data was analyzed.
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No